CLINICAL TRIAL: NCT01814865
Title: Pre-operative Assessment of the Anti-Proliferative Effects and Genomic Alterations of 2 Weeks of Abiraterone Acetate Compared to 2 Weeks of an Aromatase Inhibitor in Post-menopausal Hormone Receptor Positive Operable Breast Cancer
Brief Title: Anti-Proliferative Effects and Genomic Alterations of Abiraterone Acetate Compared to an Aromatase Inhibitor in Post-menopausal HR+ Operable Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was not acquired
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 212082BCA2004
Record Dates: First submitted 2013-03-13; First posted 2013-03-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Post-menopausal ER+ Stage I-IIIA Primary Operable Breast Cancer
Keywords: Post-menopausal; ER+; Stage I-IIIA; Operable; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Abiraterone Acetate; Prednisone; Aromatase Inhibitors; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abiraterone Acetate + Prednisone (Experimental): Abiraterone 1000mg PO OD + Prednisone 5mg PO OD x 2 weeks
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone
- Aromatase Inhibitor (Active Comparator): Anastrozole 1mg PO OD x 2 weeks
  Interventions: Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: Abiraterone Acetate — 1000 mg PO OD x 2 weeks
  Arms: Abiraterone Acetate + Prednisone
Drug: Prednisone — 5 mg PO OD x 2 weeks
  Arms: Abiraterone Acetate + Prednisone
Drug: Aromatase Inhibitor — 1 mg PO OD x 2 weeks
  Other Names: Anastrozole
  Arms: Aromatase Inhibitor

SUMMARY:
This study is being offered to patients who are post-menopausal, have breast cancer with a positive estrogen and/or progesterone hormone receptor test and are currently awaiting surgery for breast cancer.

The purpose of this study is to determine whether abiraterone acetate has different hormonal and genomic effects than non-steroidal aromatase inhibitors in the treatment of post-menopausal hormonal receptor positive primary operable breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Woman greater than or equal to 18 years of age and postmenopausal determined by one of the following:

   * bilateral surgical oophorectomy
   * age greater than or equal 60 years
   * age <60 years, with amenorrhea greater than or equal 24 months and follicle-stimulating hormone and luteinizing hormone concentrations within postmenopausal range
2. Subjects with ER+ (Allred 3-8), HER2 - primary operable T1-T3 breast cancer with a primary tumor size of ≥ 1.5 cm on physical examination or imaging studies
3. Eastern Cooperative Oncology Group (ECOG) performance status score of less than or equal to 1
4. Criterion modified per amendment 7.1 Clinical laboratory values during Screening:

   * hemoglobin greater than or equal 10.0 g/dL
   * neutrophils greater than or equal 1.5 x 109/L
   * platelets greater than or equal100 x 109/L
   * total bilirubin less than or equal to 1.5x upper limit of normal (ULN) - except for a known diagnosis of Gilbert's syndrome
   * alanine (ALT) and aspartate (AST) aminotransferase less than or equal to 1.5xULN
   * alkaline phosphatase less than or equal to 1.5xULN
   * serum creatinine <1.5xULN or creatinine clearance greater than or equal 45 mL/min
   * serum potassium greater than or equal 3.5 mM
   * serum albumin greater than or equal 3.0 g/dL
   * INR (or PT) and partial thromboplastin time (PTT) within normal limits
5. Systolic blood pressure <180 mm Hg and diastolic blood pressure <100 mm Hg [Note: Hypertension controlled by antihypertensive therapy is permitted].
6. Willing and able to adhere to prohibitions and restrictions specified in this protocol
7. Signs an informed consent document within 4 weeks before randomization indicating she understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

1. Prior treatment with ketoconazole, aminoglutethimide or a CYP17 inhibitor. [Note: Prior treatment with ketoconazole for ≤7 days is permitted and topical formulations of ketoconazole are permitted]
2. Anticancer immunotherapy, investigational agent, anticancer radiotherapy or anticancer endocrine therapy within 12 weeks before randomization
3. Use of hormone replacement therapy within the past 4 weeks
4. Serious or uncontrolled nonmalignant disease, including active or uncontrolled infection
5. Clinical or biochemical evidence of hyper-aldosteronism or hypopituitarism
6. Any condition that, in the opinion of the investigator, would compromise the well-being of the patient or that could prevent, limit, or confound the protocol-specified assessments
7. Major thoracic or abdominal surgery or significant traumatic injury with 4 weeks before randomization [Note: Patients with planned surgical procedures to be conducted under local anesthesia are not excluded from the study (e.g. intravascular device insertion)]
8. Gastrointestinal disorder interfering with study drug absorption
9. Positive serology for hepatitis B surface antigen or hepatitis C antibody
10. Active or symptomatic viral hepatitis or chronic liver disease
11. History of clinically significant heart disease, ie, myocardial infarction or arterial thrombotic event within 6 months, severe or unstable angina, or New York Heart Association Class III or IV heart disease
12. Known allergies, hypersensitivity, or intolerance to abiraterone acetate, prednisone, or their excipients
13. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before the planned first dose of study drug or is currently enrolled in an investigational study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Differences in genomic expression and biological activity | 2 weeks (baseline and day 14)
  To determine the differences in genomic expression changes with 2 weeks of abiraterone acetate plus prednisone relative to changes with 2 weeks of an aromatase inhibitor as a means to assess for potential differences in biological activity between abiraterone acetate and aromatase inhibitors in breast cancer

SECONDARY OUTCOMES:
Change in proliferation | 2 weeks (baseline and day 14)
  To compare the magnitude in change in proliferation (Ki67 as measured by IHC) with abiraterone acetate plus prednisone relative to changes in proliferation with an aromatase inhibitor following 2 weeks of pre-operative therapy
Resulting adverse events of two weeks of abiraterone acetate | 2 weeks (baseline and day 14)
  To evaluate the safety of two weeks of abiraterone acetate plus prednisone in this pre-operative population of patients.
  Safety analyses will analyze treatment-emergent adverse events coded using MedDRA resulting in death, serious adverse events, discontinuation, modification and dose interruption or day. Other safety endpoints include vital signs and clinical laboratory parameters.
Changes in plasma hormone levels | 2 weeks (baseline and day 14)
  To evaluate the changes in plasma hormone levels (androgens and estrogens) from baseline to after 2 weeks of abiraterone acetate plus prednisone

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chia, MD, Principal Investigator — British Columbia Cancer Agency
Locations (4):
- Canada (4):
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Segal Cancer Centre, Montreal, Quebec